CLINICAL TRIAL: NCT00640354
Title: Defibrillation by Automated External Defibrillators Versus Manual Defibrillators in Simulated Pediatric In-Hospital Cardiac Arrests: A Prospective Randomized Controlled Trial of Pediatric Residents
Brief Title: Time to Defibrillation Using Automated External Defibrillators by Pediatric Residents in Simulated Cardiac Arrests
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, Antonio Mott, Associate Professor, Pediatrics-Cardiology, Baylor College of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H - 18876
Record Dates: First submitted 2008-03-18; First posted 2008-03-21 (Estimated); Last update posted 2020-11-12 (Actual); Status verified 2020-11

CONDITIONS: Pediatric Residents
Keywords: Automated External Defibrillator; Resuscitation; Pediatric
MeSH Terms: interventions — Defibrillators

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Pediatric residents randomized to having an automated external defibrillator
  Interventions: Device: Automated external defibrillator
- 2 (Active Comparator): Pediatric residents randomized to having a manual defibrillator
  Interventions: Device: Manual defibrillator

INTERVENTIONS:
Device: Automated external defibrillator — Residents randomized to this group had an automated external defibrillator available for the simulated cardiac arrest. The automated external defibrillator did not actually discharge energy into the simulated patient
  Arms: 1
Device: Manual defibrillator — Residents randomized to this group had a manual defibrillator available for the simulated cardiac arrest. The defibrillator did not actually discharge energy into the simulated patient.
  Arms: 2

SUMMARY:
Automated external defibrillators have improved survival for adult in hospital cardiac arrest. Automated external defibrillators are approved for children aged 1 year and older for out of hospital cardiac arrests. It is unknown whether automated external defibrillators have a role for in hospital pediatric cardiac arrests.

The purpose of study is to compare the management of cardiac rhythm disorders by pediatric residents using an automated external defibrillator versus a standard defibrillator in simulated pediatric cardiac arrests.

It is our hypothesis that residents using an automated external defibrillator will have a shorter time to defibrillation.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric resident at Baylor College of Medicine

Exclusion Criteria:

* Not a pediatric resident at Baylor College of Medicine

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2006-12; Primary Completion 2007-02 (Actual); Study Completion 2007-02 (Actual)

PRIMARY OUTCOMES:
Time to defibrillation | Within 5 minutes of the start of the simulated cardiac arrest

CONTACTS AND LOCATIONS:
Overall Officials: Antonio R Mott, MD, Principal Investigator — Baylor College of Medicine
Locations (1):
- Texas Children's Hospital, Houston, Texas, United States

REFERENCES:
- [Background] Rossano JW, Quan L, Kenney MA, Rea TD, Atkins DL. Energy doses for treatment of out-of-hospital pediatric ventricular fibrillation. Resuscitation. 2006 Jul;70(1):80-9. doi: 10.1016/j.resuscitation.2005.10.031. Epub 2006 Jun 8. PMID 16762479
- [Background] Mogayzel C, Quan L, Graves JR, Tiedeman D, Fahrenbruch C, Herndon P. Out-of-hospital ventricular fibrillation in children and adolescents: causes and outcomes. Ann Emerg Med. 1995 Apr;25(4):484-91. doi: 10.1016/s0196-0644(95)70263-6. PMID 7710153
- [Background] Hickey RW, Cohen DM, Strausbaugh S, Dietrich AM. Pediatric patients requiring CPR in the prehospital setting. Ann Emerg Med. 1995 Apr;25(4):495-501. doi: 10.1016/s0196-0644(95)70265-2. PMID 7710155
- [Background] Samson RA, Nadkarni VM, Meaney PA, Carey SM, Berg MD, Berg RA; American Heart Association National Registry of CPR Investigators. Outcomes of in-hospital ventricular fibrillation in children. N Engl J Med. 2006 Jun 1;354(22):2328-39. doi: 10.1056/NEJMoa052917. PMID 16738269
- [Background] Samson RA, Berg RA, Bingham R; Pediatric Advanced Life Support Task Force, International Liaison Committee on Resuscitation for the American Heart Association; European Resuscitation Council. Use of automated external defibrillators for children: an update--an advisory statement from the Pediatric Advanced Life Support Task Force, International Liaison Committee on Resuscitation. Pediatrics. 2003 Jul;112(1 Pt 1):163-8. doi: 10.1542/peds.112.1.163. No abstract available. PMID 12837882
- [Background] Deakin CD, Nolan JP; European Resuscitation Council. European Resuscitation Council guidelines for resuscitation 2005. Section 3. Electrical therapies: automated external defibrillators, defibrillation, cardioversion and pacing. Resuscitation. 2005 Dec;67 Suppl 1:S25-37. doi: 10.1016/j.resuscitation.2005.10.008. No abstract available. PMID 16321714
- [Background] Larsen MP, Eisenberg MS, Cummins RO, Hallstrom AP. Predicting survival from out-of-hospital cardiac arrest: a graphic model. Ann Emerg Med. 1993 Nov;22(11):1652-8. doi: 10.1016/s0196-0644(05)81302-2. PMID 8214853
- [Background] Valenzuela TD, Roe DJ, Nichol G, Clark LL, Spaite DW, Hardman RG. Outcomes of rapid defibrillation by security officers after cardiac arrest in casinos. N Engl J Med. 2000 Oct 26;343(17):1206-9. doi: 10.1056/NEJM200010263431701. PMID 11071670
- [Background] Zafari AM, Zarter SK, Heggen V, Wilson P, Taylor RA, Reddy K, Backscheider AG, Dudley SC Jr. A program encouraging early defibrillation results in improved in-hospital resuscitation efficacy. J Am Coll Cardiol. 2004 Aug 18;44(4):846-52. doi: 10.1016/j.jacc.2004.04.054. PMID 15312869
- [Background] Gombotz H, Weh B, Mitterndorfer W, Rehak P. In-hospital cardiac resuscitation outside the ICU by nursing staff equipped with automated external defibrillators--the first 500 cases. Resuscitation. 2006 Sep;70(3):416-22. doi: 10.1016/j.resuscitation.2006.02.006. Epub 2006 Aug 14. PMID 16908093
- [Background] Woollard M, Whitfield R, Newcombe RG, Colquhoun M, Vetter N, Chamberlain D. Optimal refresher training intervals for AED and CPR skills: a randomised controlled trial. Resuscitation. 2006 Nov;71(2):237-47. doi: 10.1016/j.resuscitation.2006.04.005. Epub 2006 Sep 28. PMID 17010497
- [Derived] Rossano JW, Jefferson LS, Smith EO, Ward MA, Mott AR. Automated external defibrillators and simulated in-hospital cardiac arrests. J Pediatr. 2009 May;154(5):672-6. doi: 10.1016/j.jpeds.2008.11.051. Epub 2009 Jan 23. PMID 19167721